CLINICAL TRIAL: NCT04662710
Title: Phase 3, Randomized Study to Evaluate the Efficacy and Safety of Lenvatinib (E7080/MK-7902) Plus Pembrolizumab (MK-3475) Plus Chemotherapy Compared With Standard of Care Therapy as First-line Intervention in Participants With Advanced/Metastatic Gastroesophageal Adenocarcinoma (LEAP-015)
Brief Title: Efficacy and Safety of Lenvatinib (E7080/MK-7902) Plus Pembrolizumab (MK-3475) Plus Chemotherapy in Participants With Advanced/Metastatic Gastroesophageal Adenocarcinoma (MK-7902-015/E7080-G000-321/LEAP-015)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7902-015; MK-7902-015 (Other: MSD); E7080-G000-321 (Other: Eisai); 2051200127 (Registry Identifier: jRCT); 2023-504834-23-00 (Registry Identifier: EU CT); U1111-1288-1010 (Registry Identifier: UTN); 2020-001990-53 (EudraCT Number)
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Advanced/Metastatic Gastroesophageal Adenocarcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib; Oxaliplatin; Capecitabine; Leucovorin; Levoleucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lenvatinib + Pembrolizumab + Chemotherapy (Experimental): Participants receive lenvatinib administered orally (PO) every day (QD) in combination with pembrolizumab intravenously (IV) every 6 weeks (Q6W) plus chemotherapy with either capecitabine and oxaliplatin (CAPOX) or chemotherapy with 5-FU, leucovorin, and oxaliplatin (mFOLFOX6). Induction with lenvatinib 8 mg QD plus pembrolizumab (400 mg Q6W) plus chemotherapy (CAPOX or mFOLFOX6) will be administered for 2 cycles (approximately 12 weeks), followed by consolidation with lenvatinib 20 mg QD plus pembrolizumab (400 mg Q6W) for 16 cycles. A cycle is 6 weeks (42 days).
  Interventions: Biological: Pembrolizumab; Biological: Lenvatinib; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Leucovorin (or Levoleucovorin); Drug: 5-FU
- Chemotherapy (Experimental): Participants receive chemotherapy with either CAPOX Q3W or mFOLFOX6 Q2W. A cycle is 6 weeks (42 days).
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Leucovorin (or Levoleucovorin); Drug: 5-FU

INTERVENTIONS:
Biological: Pembrolizumab — 400 mg Q6W by IV infusion
  Other Names: MK-3475; Keytruda®
  Arms: Lenvatinib + Pembrolizumab + Chemotherapy
Biological: Lenvatinib — Administered PO QD, 8 mg induction/20 mg consolidation.
  Other Names: MK-7902; E7080
  Arms: Lenvatinib + Pembrolizumab + Chemotherapy
Drug: Oxaliplatin — 130 mg/m^2 administered by IV infusion on Day 1 of Weeks 1 and 4 of each Q6W cycle as part of CAPOX chemotherapy, or 85 mg/m^2 administered by IV infusion on Day 1 and Week 1, 3 and 5 of each Q6W cycle as part of mFOLFOX6 chemotherapy.
Drug: Capecitabine — 1000 mg/m^2 administered PO twice daily (BID) on Days 1-14, 22-35 of each Q6W cycle as part of CAPOX chemotherapy.
Drug: Leucovorin (or Levoleucovorin) — Administered by IV infusion at 400 mg/m^2 (leucovorin) or 200 mg/m^2 (levoleucovorin) on Day 1, and Week 1, 3 and 5 of each Q6W cycle as part of mFOLFOX6 chemotherapy.
Drug: 5-FU — 400 mg/m^2 bolus IV infusion followed by 2400 mg/m^2 continuous IV infusion administered on Day 1, and Week 1, 3, 5, of each Q2W cycle as part of mFOLFOX6 chemotherapy.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of lenvatinib (E7080/MK-7902) plus pembrolizumab (MK-3475) plus chemotherapy compared with chemotherapy alone in participants with advanced/metastatic gastroesophageal cancer.

The primary study hypotheses are that lenvatinib plus pembrolizumab plus chemotherapy is superior to chemotherapy alone for both overall survival (OS) and progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by blinded independent central review (BICR), in participants with programmed cell death-ligand 1 (PD-L1) Combined Positive Score (CPS) ≥1 and in all participants.

DETAILED DESCRIPTION:
There will be 2 parts to the study: a Safety Run-in (Part 1) and the Main Study (Part 2). In Part 1 (Safety Run-in), approximately 12 participants will be treated with lenvatinib in combination with pembrolizumab and chemotherapy with either capecitabine and oxaliplatin (CAPOX), or 5-fluorouracil (5-FU), Leucovorin, and oxaliplatin (mFOLFOX6). Participants will be closely followed for dose-limiting toxicities for 21 days after the first dose of study intervention.

In Part 2, up to 878 eligible participants (not including those participating in Part 1) will be randomly assigned in a 1:1 ratio to either lenvatinib plus pembrolizumab plus chemotherapy (CAPOX or mFOLFOX6) or Chemotherapy alone (CAPOX or mFOLFOX6).

Participants can receive up to 18 infusions (up to 2 years) of pembrolizumab in the first course. Participants may be eligible to receive a second course of pembrolizumab (approximately 1 year) at the investigator's discretion.

As of Amendment 8 (Effective 06/10/2025), Second Course will no longer be offered. Any participant currently receiving Second Course retreatment will be able to continue treatment as planned. Imaging will be performed per local standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically and/or cytologically confirmed diagnosis of previously untreated, locally advanced unresectable or metastatic gastroesophageal adenocarcinoma
* Is not expected to require tumor resection during the treatment course
* Has gastroesophageal adenocarcinoma that is not human epidermal growth factor receptor 2 (HER-2)/neu positive
* Has measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 by scan with IV contrast as determined by the local site investigator
* Male participants agree to refrain from donating sperm and agree to either remain abstinent from heterosexual intercourse as their preferred and usual lifestyle OR agree to use contraception, during the intervention period and for ≥7 days after last dose of lenvatinib or 90 days after last dose of chemotherapy-whichever comes last
* Female participants not pregnant or breastfeeding are eligible to participate if not a women of childbearing potential (WOCBP), or if a WOCBP they either use a contraceptive method that is highly effective OR remain abstinent from heterosexual intercourse as their preferred and usual lifestyle, and do not donate eggs (ova, oocytes) to others or freeze/store for their own use, and abstain from breastfeeding during the intervention period through 120 days after last dose of pembrolizumab, 30 days after last dose of lenvatinib, or 180 days after last dose of chemotherapy-whichever occurs last
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale within 3 days prior to the first dose of study treatment
* Has adequately controlled blood pressure with or without antihypertensive medications
* Has adequate organ function

Exclusion Criteria:

* Has had previous therapy for locally advanced unresectable or metastatic gastric/gastroesophageal junction (GEJ) esophageal adenocarcinoma
* Has had major surgery within 28 days prior to first dose of study interventions
* Has had radiotherapy within 14 days of randomization
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has severe hypersensitivity (≥Grade 3) to treatment with an monoclonal antibody (mAb) or known sensitivity or intolerance to any component of lenvatinib, pembrolizumab, study chemotherapy agents and/or to any excipients, murine proteins, or platinum containing products
* Has had an allogeneic tissue/solid organ transplant
* Has perforation risks or significant gastrointestinal (GI) bleeding
* Has GI obstruction, poor oral intake (CAPOX participants), or difficulty in taking oral medication (CAPOX participants)
* Has received prior therapy with an anti-programmed cell death 1 (PD-1), anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor
* Has received prior therapy with anti- vascular endothelial growth factor (VEGF) tyrosine kinase inhibitor or anti-VEGF mAb
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study drug
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs)
* Has radiographic evidence of encasement or invasion of a major blood vessel, or of intratumoral cavitation
* Has inadequate cardiac function
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has poorly controlled diarrhea
* Has accumulation of pleural, ascitic, or pericardial fluid requiring drainage or diuretic drugs within 2 weeks prior to enrollment
* Has peripheral neuropathy ≥Grade 2
* Has a known history of human immunodeficiency virus (HIV) or HIV 1/2 antibodies
* Has a known history of hepatitis B (defined as HBsAg reactive) or known active hepatitis C virus (defined as HCV ribonucleic acid (RNA) [qualitative] is detected) infection
* Has weight loss of >20% within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 895 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (177):
- United States (12):
  - UCLA Hematology/Oncology - Santa Monica ( Site 0003), Los Angeles, California
  - Georgetown University Medical Center ( Site 0009), Washington D.C., District of Columbia
  - James Graham Brown Cancer Center ( Site 0017), Louisville, Kentucky
  - Johns Hopkins University ( Site 0052), Baltimore, Maryland
  - Dana Farber Cancer Center ( Site 0019), Boston, Massachusetts
  - UMASS Memorial Medical Center ( Site 0020), Worcester, Massachusetts
  - Henry Ford Health System ( Site 0023), Detroit, Michigan
  - Cancer and Hematology Centers of Western Michigan ( Site 0025), Grand Rapids, Michigan
  - Washington University School of Medicine ( Site 0027), St Louis, Missouri
  - Mount Sinai Hospital ( Site 0051), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 0032), New York, New York
  - AHN West Penn Hospital-AHN Esophageal and Lung Institute ( Site 0058), Pittsburgh, Pennsylvania
- Argentina (7):
  - IDIM Instituto de Diagnostico e Investigaciones Metabolicas ( Site 0202), Caba, Buenos Aires
  - Instituto Medico Alexander Fleming ( Site 0208), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Fundacion Favaloro ( Site 0201), Buenos Aires
  - Hospital Aleman ( Site 0210), Buenos Aires
  - Hospital Municipal de Gastroenterologia Dr. Bonorino Udaondo ( Site 0207), Buenos Aires
  - CEMIC ( Site 0209), Buenos Aires
  - Hospital Privado de Cordoba ( Site 0204), Córdoba
- Australia (4):
  - Nepean Hospital ( Site 2305), Kingswood, New South Wales
  - Wollongong Hospital ( Site 2307), Wollongong, New South Wales
  - Royal Brisbane and Women s Hospital ( Site 2304), Herston, Queensland
  - Hollywood Private Hospital-Medical Oncology ( Site 2308), Nedlands, Western Australia
- Belgium (4):
  - CHU UCL Namur Site de Godinne ( Site 1005), Yvoir, Namur
  - UZ Gent ( Site 1002), Ghent, Oost-Vlaanderen
  - UZ Leuven ( Site 1004), Leuven, Vlaams-Brabant
  - AZ Delta ( Site 1006), Roeselare, West-Vlaanderen
- Canada (3):
  - Queen Elizabeth II Health Sciences Centre ( Site 0101), Halifax, Nova Scotia
  - Hamilton Health Sciences - Juravinski Site ( Site 0106), Hamilton, Ontario
  - CIUSSS de l Estrie - CHUS - Centre Hosp. Univ. Sherbrooke ( Site 0103), Sherbrooke, Quebec
- Chile (6):
  - IC La Serena Research ( Site 0410), La Serena, Coquimbo Region
  - Clinica Universidad Catolica del Maule ( Site 0411), Talca, Maule Region
  - Fundacion Arturo Lopez Perez FALP ( Site 0403), Santiago, Region M. de Santiago
  - Clínica San Carlos de Apoquindo Red Salud UC Christus ( Site 0407), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0404), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 0414), Temuco, Región de la Araucanía
- China (28):
  - Anhui Provincial Hospital ( Site 2415), Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences ( Site 2403), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 2453), Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital ( Site 2408), Fuzhou, Fujian
  - The 900th Hospital of the Joint Logistics Support Force of the Chinese People's Liberation Army ( Si, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University ( Site 2420), Xiamen, Fujian
  - The First Affiliated Hospital of Xiamen University ( Site 2446), Xiamen, Fujian
  - Zhongshan Hospital Affiliated to Xiamen University ( Site 2421), Xiamen, Fujian
  - First Hospital of Lanzhou University ( Site 2417), Lanzhou, Gansu
  - Nanfang Hospital ( Site 2456), Guangzhou, Guangdong
  - The Affiliated Hospital Of Hainan Medical University-Cancer rehabilitation and palliative treatment, Haikou, Hainan
  - Fourth Hospital Of Hebei Medical University ( Site 2441), Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital ( Site 2410), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 2443), Zhengzhou, Henan
  - Hubei Cancer Hospital ( Site 2429), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 2440), Changsha, Hunan
  - Changzhou Cancer Hospital-Department of Oncology ( Site 2458), Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital ( Site 2419), Nanjing, Jiangsu
  - Nantong Tumor Hospital-Digestive Oncology ( Site 2464), Nantong, Jiangsu
  - Jilin Cancer Hospital ( Site 2438), Changchun, Jilin
  - Tang Du Hospital ( Site 2432), Xi'an, Shaanxi
  - LinYi Cancer Hospital-Gastrology department ( Site 2463), Linyi, Shandong
  - Shanghai General Hospital ( Site 2424), Shanghai, Shanghai Municipality
  - Shanghai East Hospital ( Site 2455), Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute & Hospital ( Site 2447), Tianjin, Tianjin Municipality
  - Cancer Hospital Affiliated to Xinjiang Medical University ( Site 2428), Ürümqi, Xinjiang
  - The First Affiliated Hospital of Zhejiang University ( Site 2414), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital ( Site 2412), Hangzhou, Zhejiang
- Colombia (6):
  - Clinica de la Costa S.A.S. ( Site 0502), Barranquilla, Atlántico
  - Clinica Colsanitas S.A. Sede Clinica Universitaria Colombia ( Site 0501), Bogotá, Bogota D.C.
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 0508), Valledupar, Cesar Department
  - Oncomedica S.A. ( Site 0507), Montería, Departamento de Córdoba
  - Instituto Cancerologico de Narino Ltda ( Site 0504), Pasto, Departamento de Nariño
  - Oncologos del Occidente S.A. ( Site 0525), Pereira, Risaralda Department
- Costa Rica (2):
  - CIMCA-Hemato-Oncology ( Site 0601), San José, Provincia de San José
  - Hospital Metropolitano - Sede Lindora-Metropolitano Research Institute Sede Lindora ( Site 0602), Santa Ana, Provincia de San José
- France (10):
  - Hôpital Edouard Herriot ( Site 1116), Lyon, Auvergne-Rhône-Alpes
  - Centre Francois Baclesse ( Site 1107), Caen, Calvados
  - Centre Georges Francois Leclerc ( Site 1106), Dijon, Cote-d Or
  - CHU Bordeaux Haut-Leveque ( Site 1110), Pessac, Gironde
  - Centre Hospitalier Annecy Genevois ( Site 1117), Epagny Metz-Tessy, Haute-Savoie
  - CHU Hotel Dieu Nantes ( Site 1101), Nantes, Pays de la Loire Region
  - Hopital Henri Mondor ( Site 1105), Créteil, Val-de-Marne
  - Institut du Cancer Avignon-Provence ( Site 1103), Avignon, Vaucluse
  - Hopital Saint Louis ( Site 1100), Paris
  - CHU Hopital Saint Antoine ( Site 1102), Paris
- Germany (7):
  - Klinikum Rechts der Isar der TU Muenchen ( Site 1200), Muechen, Bavaria
  - Universitaetsklinikum Regensburg ( Site 1203), Regensburg, Bavaria
  - Krankenhaus Nordwest ( Site 1205), Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover ( Site 1210), Hanover, Lower Saxony
  - Universitaetsklinikum Leipzig ( Site 1211), Leipzig, Saxony
  - Charite Berlin Campus Virchow-Klinikum ( Site 1202), Berlin
  - Facharztzentrum Eppendorf ( Site 1201), Hamburg
- Guatemala (6):
  - Clinica Privada Dr Rixci Ramirez Fallas ( Site 0702), Guatemala City
  - Oncologika S.A. ( Site 0704), Guatemala City
  - Oncomedica ( Site 0701), Guatemala City
  - Soluciones Gastrointestinales S.A. ( Site 0706), Guatemala City
  - Sanatorio Nuestra Senora del Pilar ( Site 0705), Guatemala City
  - Medi-K Cayala ( Site 0700), Guatemala City
- Hong Kong (3):
  - Prince of Wales Hospital ( Site 2503), Hong Kong
  - Princess Margaret Hospital. ( Site 2502), Hong Kong
  - Queen Mary Hospital ( Site 2501), Hong Kong
- Ireland (2):
  - St James Hospital ( Site 1400), Dublin, Leinster
  - Beaumont Hospital ( Site 1402), Dublin
- Israel (7):
  - Soroka Medical Center ( Site 1507), Beersheba
  - Hillel Yaffe Medical Center ( Site 1503), Hadera
  - Rambam Health Care Campus-Oncology Division ( Site 1502), Haifa
  - Hadassah Ein Kerem Medical Center ( Site 1501), Jerusalem
  - Meir Medical Center ( Site 1504), Kfar Saba
  - Rabin Medical Center ( Site 1506), Petah Tikva
  - Sourasky Medical Center ( Site 1500), Tel Aviv
- Italy (8):
  - Istituto Scientifico Romagnolo per Studio e Cura Tumori IRST ( Site 1608), Meldola, Abruzzo
  - Presidio Ospedaliero Universitario Santa Maria della Misericordia ( Site 1609), Udine, Friuli Venezia Giulia
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1610), Milan, Lombardy
  - Humanitas Research Hospital ( Site 1600), Rozzano, Lombardy
  - AULSS8 Berica-Ospedale S.Bortolo ( Site 1607), Vicenza, Veneto
  - Azienda Ospedaliera Mater Domini-Translational Oncology Unit ( Site 1611), Catanzaro
  - IRCCS Ospedale San Raffaele di Milano ( Site 1603), Milan
  - A.O.U. Universita degli Studi della Campania-Luigi Vanvitelli ( Site 1604), Napoli
- Japan (16):
  - Aichi Cancer Center Hospital ( Site 2603), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 2601), Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 2610), Matsuyama, Ehime
  - Hyogo Cancer Center ( Site 2621), Akashi, Hyōgo
  - Kobe City Medical Center General Hospital ( Site 2606), Kobe, Hyōgo
  - Ibaraki Prefectural Central Hospital ( Site 2618), Kasama, Ibaraki
  - Kagawa University Hospital ( Site 2611), Kita-gun, Kagawa-ken
  - Kanagawa Cancer Center ( Site 2608), Yokohama, Kanagawa
  - Kansai Medical University Hospital ( Site 2622), Hirakata, Osaka
  - Kindai University Hospital ( Site 2600), Sayama, Osaka
  - Saitama Cancer Center ( Site 2604), Kitaadachi-gun, Saitama
  - National Hospital Organization Kyushu Cancer Center ( Site 2609), Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital ( Site 2612), Hiroshima
  - Osaka International Cancer Institute ( Site 2607), Osaka
  - National Cancer Center Hospital ( Site 2602), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 2605), Tokyo
- Poland (5):
  - Przychodnia Lekarska KOMED ( Site 1701), Konin, Greater Poland Voivodeship
  - Szpital Kliniczny im. Heliodora Swiecickiego Uniwers Medyczn ( Site 1703), Poznan, Greater Poland Voivodeship
  - Dolnoslaskie Centrum Onkologii. ( Site 1712), Wroclaw, Lower Silesian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 1704), Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 1702), Przemyśl, Podkarpackie Voivodeship
- Russia (9):
  - Chelyabinsk Regional Clinical Oncological Dispensary ( Site 1816), Chelyabinsk, Chelyabinsk Oblast
  - National Medical and Surgical Center n.a.N.I.Pirogov ( Site 1805), Moscow, Moscow
  - Blokhin National Medical Oncology ( Site 1800), Moscow, Moscow
  - Central Clinical Hospital with Polyclinic ( Site 1801), Moscow, Moscow
  - Medical University REAVIZ ( Site 1814), Samara, Samara Oblast
  - Leningrad Regional Oncology Center ( Site 1810), Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 1809), Saint Petersburg, Sankt-Peterburg
  - St Petersburg City Clinical Oncology Dispensary ( Site 1808), Saint Petersburg, Sankt-Peterburg
  - Yaroslavl Regional SBIH Clinical Oncology Hospital ( Site 1821), Yaroslavl, Yaroslavl Oblast
- South Korea (9):
  - Hallym University Sacred Heart Hospital ( Site 2806), Anyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 2804), Seongnam-si, Kyonggi-do
  - Asan Medical Center ( Site 2802), Songpagu, Seoul
  - Konyang University ( Site 2807), Daejeon, Taejon-Kwangyokshi
  - Seoul National University Hospital ( Site 2803), Seoul
  - Severance Hospital Yonsei University Health System ( Site 2800), Seoul
  - Gangnam Severance Hospital ( Site 2805), Seoul
  - Samsung Medical Center ( Site 2801), Seoul
  - Korea University Guro Hospital ( Site 2808), Seoul
- Spain (4):
  - Hospital Universitario Marques de Valdecilla ( Site 1902), Santander, Cantabria
  - Hospital Universitario General de Asturias ( Site 1901), Oviedo, Principality of Asturias
  - Hospital General Universitari Vall d Hebron ( Site 1907), Barcelona
  - Hospital General Gregorio Maranon de Madrid ( Site 1904), Madrid
- Taiwan (4):
  - China Medical University Hospital ( Site 2903), Taichung
  - National Cheng Kung University Hospital ( Site 2904), Tainan
  - National Taiwan University Hospital ( Site 2901), Taipei
  - Chang Gung Medical Foundation. Linkou ( Site 2902), Taoyuan District
- Turkey (Türkiye) (7):
  - Sakarya Universitesi Tip Fakultesi ( Site 2007), Sakarya, Istanbul
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 2003), Ankara
  - Memorial Ankara Hastanesi ( Site 2004), Ankara
  - Trakya Universitesi Tip Fakultesi ( Site 2000), Edirne
  - Ataturk Universitesi Tip Fakultesi Hastanesi ( Site 2005), Erzurum
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 2002), Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi ( Site 2001), Izmir
- United Kingdom (8):
  - Addenbrooke's Hospital ( Site 2200), Cambridge, Cambridgeshire
  - Ninewells Hospital and Medical School ( Site 2207), Dundee, Dundee City
  - The Beatson West of Scotland Cancer Centre ( Site 2204), Glasgow, Glasgow City
  - University College London Hospitals NHS Foundation Trust ( Site 2201), London, London, City of
  - Royal Marsden NHS Foundation Trust ( Site 2202), London, London, City of
  - Royal Marsden NHS Trust ( Site 2203), Sutton, Surrey
  - University Hospital Coventry and Warwickshire NHS Trust ( Site 2205), Coventry, Warwickshire
  - The Christie NHS Foundation Trust ( Site 2209), Manchester

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Shitara K, Lorenzen S, Li J, Bai Y, Fernandez MG, Aguilar M, Shoji H, Reyes-Cosmelli F, Pena YR, Corrales L, Wyrwicz L, Eyzaguirre DA, Pan Y, Ryu MH, Cohen DJ, Wainberg ZA, Ku G, Tabernero J, Van Cutsem E, Qin SK, Oh DY, Xu J, Liang LW, Bordia S, Bhagia P, Rha SY; LEAP-015 Investigators. Lenvatinib Plus Pembrolizumab and Chemotherapy Versus Chemotherapy in Advanced Metastatic Gastroesophageal Adenocarcinoma: The Phase III, Randomized LEAP-015 Study. J Clin Oncol. 2025 Aug;43(22):2502-2514. doi: 10.1200/JCO-25-00748. Epub 2025 May 31. PMID 40448579
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26248&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included 2 parts: Part 1 was an open-label, safety run-in to evaluate the safety and tolerability of treatment with pembrolizumab + lenvatinib + chemotherapy. Participants in Part 1 continued to receive study intervention and were followed in the posttreatment period as applicable. Part 2 (main study) evaluated safety and efficacy. Participants were randomized to receive either treatment with pembrolizumab + lenvatinib + chemotherapy, or chemotherapy only.
Groups:
- Part 1 : Lenvatinib + Pembrolizumab + Chemotherapy; Part 2: Lenvatinib + Pembrolizumab + Chemotherapy: Participants received lenvatinib administered orally (PO) every day (QD) in combination with pembrolizumab intravenously (IV) every 6 weeks (Q6W) plus chemotherapy with either capecitabine and oxaliplatin (CAPOX) or chemotherapy with 5-FU, leucovorin, and oxaliplatin (mFOLFOX6). Induction with lenvatinib 8 mg QD plus pembrolizumab plus chemotherapy (CAPOX or mFOLFOX6) was administered for 2 cycles, followed by consolidation with lenvatinib 20 mg QD plus pembrolizumab for up to 16 cycles. A cycle is 6 weeks (42 days).
- Part 2: Chemotherapy: Participants received chemotherapy with either CAPOX every 3 weeks (Q3W) or mFOLFOX6 every 2 weeks (Q2W).
Period: Overall Study
Arm/Group | Part 1 : Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Chemotherapy
Started | 15 | 443 | 437
Treated | 15 | 441 | 429
Received Second Course of Pembrolizumab +/- Lenvatinib | 1 | 3 | 0
Completed | 0 | 0 | 0
Not Completed | 15 | 443 | 437
Not completed — Death | 14 | 331 | 367
Not completed — Ongoing | 1 | 109 | 56
Not completed — Withdrawal by Subject | 0 | 3 | 14

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Lenvatinib +Pembrolizumab + Chemotherapy; Part 2: Lenvatinib + Pembrolizumab + Chemotherapy: Participants received lenvatinib administered orally QD in combination with IV pembrolizumab Q6W plus chemotherapy with either CAPOX or chemotherapy with mFOLFOX6. Induction with lenvatinib 8 mg QD plus pembrolizumab (plus chemotherapy (CAPOX or mFOLFOX6) was administered for 2 cycles, followed by consolidation with lenvatinib 20 mg QD plus pembrolizumab for up to 16 cycles. A cycle is 6 weeks (42 days).
- Part 2: Chemotherapy: Participants received chemotherapy with either CAPOX Q3W or mFOLFOX6 Q2W.
- Total: Total of all reporting groups
Arm/Group | Part 1: Lenvatinib +Pembrolizumab + Chemotherapy | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Chemotherapy | Total
Number analyzed (Participants) | 15 | 443 | 437 | 895
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.9 (59.7) | 59.7 (12.5) | 59.1 (12.0) | 59.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 151 | 131 | 290
  Male | 7 | 292 | 306 | 605
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 116 | 115 | 238
  Not Hispanic or Latino | 8 | 319 | 313 | 640
  Unknown or Not Reported | 0 | 8 | 9 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 11 | 15 | 26
  Asian | 4 | 164 | 161 | 329
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 11 | 235 | 223 | 469
  More than one race | 0 | 30 | 36 | 66
  Unknown or Not Reported | 0 | 2 | 1 | 3
Geographic Region of Enrolling Site [Count of Participants; unit: Participants] — Participants were classified according to the geographic region of enrolling site in the following categories: East Asia, North America + Western Europe (included United States, Canada, Belgium, France, Germany, Ireland, Italy, Spain, United Kingdom, Israel and Australia) and Rest of World.
  Participants
    East Asia | 4 | 161 | 160 | 325
    North America + Western Europe | 5 | 125 | 122 | 252
    Rest of the World | 6 | 157 | 155 | 318
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Participants were assessed for ECOG performance status: Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature.
  Participants
    ECOG 0 | 11 | 204 | 204 | 419
    ECOG 1 | 4 | 239 | 233 | 476
Intended Chemotherapy [Count of Participants; unit: Participants] — Participants were classified according to the type of chemotherapy they were intended to receive: CAPOX [capecitabine 1000 mg/m2 BID for 14 days (oral) and oxaliplatin 130 mg/m2 (IV) q3w] or mFOLFOX6 [oxaliplatin 85 mg/m2 (IV), 5-FU 400 mg/m2 (bolus IV)plus 2400 mg/m2 (continuous IV), and leucovorin 400mg/m2 (IV) or levoleucovorin 200 mg/m2 (IV) q2w]
  Participants
    CAPOX | 7 | 232 | 225 | 464
    mFOLFOX6 | 8 | 209 | 204 | 421
    Missing | 0 | 2 | 8 | 10

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as a specific adverse event graded for toxicity using the Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Hematologic DLTs included Grade 4 neutropenia lasting for ≥7 days, Grade 3 or Grade 4 febrile neutropenia, Grade 3 thrombocytopenia with bleeding, Grade 4 thrombocytopenia, or Grade 4 anemia. Nonhematologic DLTs included any other Grade 4 or Grade 5 toxicity, Grade 3 toxicities lasting >3 days (excluding nausea, vomiting, and diarrhea controlled by medical intervention within 72 hours, and Grade 3 rash in the absence of desquamation with no mucosal involvement), Grade 3 hypertension not able to be controlled by medication, ≥ Grade 3 gastrointestinal perforation, ≥Grade 3 wound dehiscence requiring medical or surgical intervention, any grade thromboembolic event, or any Grade 3 nonhematologic laboratory value if medical intervention was required or the abnormality led to hospitalization. The number of participants in Part 1 with DLTs is reported.
Time Frame: Up to ~21 days
Population: All randomized participants who received at least 1 dose of study intervention. Per protocol, only participants in part 1 were included
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 : Lenvatinib + Pembrolizumab + Chemotherapy: Participants received lenvatinib administered orally QD in combination with IV pembrolizumab Q6W plus chemotherapy with either CAPOX or chemotherapy with mFOLFOX6. Induction with lenvatinib 8 mg QD plus pembrolizumab plus chemotherapy (CAPOX or mFOLFOX6) was administered for 2 cycles, followed by consolidation with lenvatinib 20 mg QD plus pembrolizumab for up to 16 cycles. A cycle is 6 weeks (42 days).
Arm/Group | Part 1 : Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Chemotherapy
Number analyzed (Participants) | 15 | 0 | 0
Participants | 2 |  |

2. Primary Outcome: Part 1: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants in Part 1 with AEs is reported
Time Frame: Up to ~44 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Safety Run-In: Lenvatinib + Pembrolizumab + Chemotherapy: Participants received lenvatinib administered orally QD in combination with IV pembrolizumab Q6W plus chemotherapy with either CAPOX or chemotherapy with mFOLFOX6.
Arm/Group | Safety Run-In: Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Chemotherapy
Number analyzed (Participants) | 15 | 0 | 0
Participants | 15 |  |

3. Primary Outcome: Part 1: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants in Part 1 that discontinued study treatment due to an AE is reported.
Time Frame: Up to ~29 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run-In: Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Chemotherapy
Number analyzed (Participants) | 15 | 0 | 0
Participants | 5 |  |

4. Primary Outcome: Part 2: Overall Survival (OS) in Participants With Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥1
Description: OS is defined as the time from randomization to death due to any cause. OS is reported by treatment arm for PD-L1 CPS ≥1 participants in Part 2.
Time Frame: Up to ~41 months
Population: All randomized participants, whether or not study intervention was administered, with PD-L1 CPS≥1 and who had available data for the outcome measure at the time of final analysis. Per protocol, participants in part 1 of the study were not included in the OS analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Chemotherapy
Number analyzed (Participants) | 334 | 355
Months | 12.6 [10.6 to 14.2] | 12.9 [11.6 to 14.6]
Statistical Analysis 1: Comparison: Part 2: Lenvatinib + Pembrolizumab + Chemotherapy vs Part 2: Chemotherapy; Test type: Superiority; p = .0244, Log Rank — One-sided p-value based on log-rank test stratified by region, ECOG performance status, and chemotherapy type; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.71 to 1.00] — HR based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by region, ECOG performance status, and chemotherapy type

5. Primary Outcome: Part 2: OS in All Participants
Description: OS is defined as the time from randomization to death due to any cause. OS is reported by treatment arm for all participants in Part 2.
Time Frame: Up to ~41 months
Population: All randomized participants, whether or not study intervention was administered and who had available data for the outcome measure at the time of final analysis. Per protocol, participants in part 1 of the study were not included in the OS analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Chemotherapy
Number analyzed (Participants) | 443 | 437
Months | 13.1 [11.6 to 14.3] | 13.0 [11.6 to 14.7]
Statistical Analysis 1: Comparison: Part 2: Lenvatinib + Pembrolizumab + Chemotherapy vs Part 2: Chemotherapy; Test type: Superiority; p = 0.0330, Log Rank — One-sided p-value based on log-rank test stratified by region, ECOG performance status and chemotherapy type; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.75 to 1.01] — HR based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by region, ECOG performance status, and chemotherapy

6. Primary Outcome: Part 2: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) in Participants With PD-L1 CPS ≥1
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 by BICR or death from any cause, whichever occurs first. Per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. PFS is reported by treatment arm for PD-L1 CPS ≥1 participants in Part 2.
Time Frame: Up to ~29 months
Population: All randomized participants, whether or not study intervention was administered, with PD-L1 CPS ≥1 and who had available data for the outcome measure at the time of final analysis. Per protocol, participants in part 1 of the study were not included in the PFS analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Chemotherapy
Number analyzed (Participants) | 333 | 355
Months | 7.3 [6.8 to 8.3] | 6.9 [5.8 to 7.2]
Statistical Analysis 1: Comparison: Part 2: Lenvatinib + Pembrolizumab + Chemotherapy vs Part 2: Chemotherapy; Test type: Superiority; p = .0012, Log Rank — One-sided p-value based on log-rank test stratified by region, performance status, and chemotherapy type; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.62 to 0.90] — [estimate comment as in outcome 4, analysis 1]

7. Primary Outcome: Part 2: PFS Per RECIST 1.1 as Assessed by BICR in All Participants
Description: PFS is defined as the time from randomization to the first documented PD per RECIST 1.1 by BICR or death from any cause, whichever occurs first. Per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. PFS is reported by treatment arm for all participants in Part 2.
Time Frame: Up to ~29 months
Population: All randomized participants, whether or not study intervention was administered and who had available data for the outcome measure at the time of final analysis. Per protocol, participants in part 1 of the study were not included in the PFS analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Chemotherapy
Number analyzed (Participants) | 443 | 437
Months | 7.2 [6.8 to 8.3] | 7.0 [6.4 to 7.5]
Statistical Analysis 1: Comparison: Part 2: Lenvatinib + Pembrolizumab + Chemotherapy vs Part 2: Chemotherapy; Test type: Superiority; p = 0.0019, Log Rank — One-sided p-value based on log-rank test stratified by region, ECOG performance status, and chemotherapy type; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.66 to 0.92] — [estimate comment as in outcome 4, analysis 1]

8. Secondary Outcome: Part 2: Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by BICR in Participants With PD-L1 CPS ≥1
Description: ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, and assessed by BICR. ORR is reported by treatment arm for PD-L1 CPS ≥1 participants in Part 2.
Time Frame: Up to ~29 months
Population: All randomized participants, whether or not study intervention was administered, with PD-L1 CPS ≥1 and who had available data for the outcome measure at the time of final analysis. Per protocol, participants in part 1 of the study were not included in the ORR analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Chemotherapy
Number analyzed (Participants) | 333 | 355
Percentage of Participants | 59.5 [54.0 to 64.8] | 45.4 [40.1 to 50.7]
Statistical Analysis 1: Comparison: Part 2: Lenvatinib + Pembrolizumab + Chemotherapy vs Part 2: Chemotherapy; ORR comparison between groups is based on Miettinen & Nurminen method stratified by region, ECOG performance status, and type of chemotherapy; Test type: Superiority; p < 0.0001, t-test, 1 sided; Difference in Percentage = 14.3, 95% CI 2-sided [6.9 to 21.5]

9. Secondary Outcome: Part 2: ORR Per RECIST 1.1 as Assessed by BICR in All Participants
Description: ORR is defined as the percentage of participants in the analysis population who have a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, and assessed by BICR. ORR is reported by treatment arm for all participants in Part 2.
Time Frame: Up to ~29 months
Population: All randomized participants, whether or not study intervention was administered and who had available data for the outcome measure at the time of final analysis. Per protocol, participants in part 1 of the study were not included in the ORR analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Chemotherapy
Number analyzed (Participants) | 443 | 437
Percentage of Participants | 58.0 [53.3 to 62.7] | 43.9 [39.2 to 48.7]
Statistical Analysis 1: Comparison: Part 2: Lenvatinib + Pembrolizumab + Chemotherapy vs Part 2: Chemotherapy; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.0001, t-test, 1 sided; Difference in Percentage = 14.2, 95% CI 2-sided [7.7 to 20.6]

10. Secondary Outcome: Part 2: Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR in Participants With PD-L1 CPS ≥1
Description: For participants who demonstrated confirmed CR or PR, DOR is defined as the time from the first CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) to subsequent PD or death due to any cause, whichever occurs first. Per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR is reported by treatment arm for PD-L1 CPS ≥1 participants in Part 2.
Time Frame: Up to ~41 months
Population: All randomized participants who achieved CR or PR with PD-L1 CPS > or =1 and who had available data for the outcome measure at the time of final analysis. Participants were analyzed in the treatment group to which they were randomized. Per protocol, participants in part 1 of the study were not included in the DOR analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Chemotherapy
Number analyzed (Participants) | 198 | 161
Months | 8.5 [7.1 to 12.5] | 6.5 [5.6 to 7.0]

11. Secondary Outcome: Part 2: DOR Per RECIST 1.1 as Assessed by BICR in All Participants
Description: For participants who demonstrated confirmed CR or PR, DOR is defined as the time from the first CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) to subsequent PD or death due to any cause, whichever occurs first. Per RECIST 1.1 modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR is reported by treatment arm for all participants in Part 2.
Time Frame: Up to ~41 months
Population: All randomized participants who achieved CR or PR and who had available data for the outcome measure at the time of final analysis. Participants were analyzed in the treatment group to which they were randomized. Per protocol, participants in part 1 of the study were not included in the DOR analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy | Part 2: Chemotherapy
Number analyzed (Participants) | 255 | 192
Months | 8.6 [7.3 to 12.4] | 6.7 [5.6 to 7.7]

12. Secondary Outcome: Part 2: Number of Participants With AEs
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants in Part 2 with AEs is reported by treatment arm.
Time Frame: Up to ~41 months
Reporting Status: Not Posted, anticipated posting 2027-03

13. Secondary Outcome: Part 2: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants in Part 2 that discontinued study treatment due to an AE is reported by treatment arm.
Time Frame: Up to ~41 months
Reporting Status: Not Posted, anticipated posting 2027-03

ADVERSE EVENTS:
Time Frame: Up to approximately 44 months
Description: All cause-mortality includes all randomized participants, whether or not study intervention was administered. The SAE and other adverse events population includes all randomized participants who received at least 1 dose of study intervention. Per protocol, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to the drug are excluded.
Groups:
- Part 1: Lenvatinib + Pembrolizumab + Chemotherapy First Course: Participants received lenvatinib administered orally QD in combination with IV pembrolizumab Q6W plus chemotherapy with either CAPOX or chemotherapy with mFOLFOX6. Induction with lenvatinib 8 mg QD plus pembrolizumab plus chemotherapy (CAPOX or mFOLFOX6) was administered for 2 cycles, followed by consolidation with lenvatinib 20 mg QD plus pembrolizumab for up to 16 cycles. A cycle is 6 weeks (42 days).
- Part 2: Lenvatinib + Pembrolizumab + Chemotherapy First Course: Participants received lenvatinib administered orally QD in combination with IV pembrolizumab Q6W plus chemotherapy with either CAPOX or chemotherapy with mFOLFOX6. Induction with lenvatinib 8 mg QD plus pembrolizumab (plus chemotherapy (CAPOX or mFOLFOX6) was administered for 2 cycles, followed by consolidation with lenvatinib 20 mg QD plus pembrolizumab for up to 16 cycles. A cycle is 6 weeks (42 days).
- Chemotherapy First Course: Participants received chemotherapy with either CAPOX Q3W or mFOLFOX6 Q2W. A cycle is 6 weeks (42 days).
- Part 1: Pembrolizumab +/-Lenvatinib Second Course: Participants treated with pembrolizumab who completed 18 cycles of treatment with SD or better, or participants who attained an investigator-determined CR and received at least 4 cycles of pembrolizumab were eligible for retreatment with up to an additional 9 cycles of pembrolizumab if they experienced radiographic disease progression confirmed by BICR after stopping treatment in the initial treatment phase. Lenvatinib was administered per investigator's discretion
- Part 2: Pembrolizumab +/-Lenvatinib Second Course: Participants treated with pembrolizumab who completed 18 cycles of treatment with SD or better, or participants who attained an investigator-determined CR and received at least 4 cycles of pembrolizumab were eligible for retreatment with up to an additional 9 cycles of pembrolizumab if they experience radiographic disease progression confirmed by BICR after stopping treatment in the initial treatment phase. Lenvatinib was administered per investigator's discretion
Arm/Group | Part 1: Lenvatinib + Pembrolizumab + Chemotherapy First Course | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy First Course | Chemotherapy First Course | Part 1: Pembrolizumab +/-Lenvatinib Second Course | Part 2: Pembrolizumab +/-Lenvatinib Second Course
All-Cause Mortality (participants affected / at risk) | 13/15 | 333/443 | 374/437 | 1/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 6/15 | 226/441 | 137/429 | 0/1 | 1/3
Other Adverse Events (participants affected / at risk) | 14/15 | 435/441 | 406/429 | 0/1 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Lenvatinib + Pembrolizumab + Chemotherapy First Course (N=15) | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy First Course (N=441) | Chemotherapy First Course (N=429) | Part 1: Pembrolizumab +/-Lenvatinib Second Course (N=1) | Part 2: Pembrolizumab +/-Lenvatinib Second Course (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (6) | 2 (2) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dihydropyrimidine dehydrogenase deficiency (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 13 (14) | 4 (4) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 6 (7) | 4 (4) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (4) | 6 (8) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3) | 11 (12) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 6 (6) | 2 (2) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 3 (6) | 4 (4) | 0 (0) | 0 (0)
Oesophageal food impaction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 9 (9) | 9 (9) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 10 (12) | 7 (7) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Medical device pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 4 (4) | 4 (4) | 0 (0) | 0 (0)
Vascular device occlusion (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholangitis sclerosing (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematological infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 4 (5) | 10 (11) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis chemical (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 4 (4) | 10 (11) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vagus nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Immune-mediated nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7) | 9 (9) | 0 (0) | 0 (0)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Lenvatinib + Pembrolizumab + Chemotherapy First Course (N=15) | Part 2: Lenvatinib + Pembrolizumab + Chemotherapy First Course (N=441) | Chemotherapy First Course (N=429) | Part 1: Pembrolizumab +/-Lenvatinib Second Course (N=1) | Part 2: Pembrolizumab +/-Lenvatinib Second Course (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 159 (249) | 161 (241) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 10 (11) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 31 (31) | 7 (8) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 4 (4) | 127 (139) | 5 (5) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 25 (27) | 18 (23) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 90 (110) | 71 (86) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 36 (39) | 21 (30) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 15 (17) | 22 (24) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 104 (130) | 88 (115) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (11) | 201 (339) | 123 (192) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 29 (30) | 7 (7) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 22 (25) | 19 (22) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 27 (27) | 20 (23) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 10 (11) | 11 (13) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (14) | 196 (290) | 193 (295) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 69 (75) | 40 (49) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (14) | 110 (166) | 105 (147) | 0 (0) | 0 (0)
Asthenia (General disorders) | 5 (6) | 74 (92) | 69 (100) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (4) | 129 (162) | 79 (104) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 2 (4) | 51 (62) | 26 (30) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 30 (36) | 25 (28) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 59 (83) | 36 (55) | 0 (0) | 0 (0)
Temperature intolerance (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 1 (1) | 12 (13) | 11 (13) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 10 (11) | 4 (4) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 5 (5) | 10 (12) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 45 (48) | 43 (44) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 2 (3) | 2 (2) | 2 (4) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 32 (51) | 13 (16) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (4) | 94 (128) | 76 (126) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 2 (2) | 55 (85) | 38 (56) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 109 (159) | 102 (162) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 2 (2) | 19 (30) | 15 (23) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 33 (41) | 44 (50) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (3) | 52 (86) | 48 (77) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 7 (8) | 7 (12) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 32 (39) | 7 (8) | 0 (0) | 0 (0)
Blood folate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 2 (4) | 7 (15) | 11 (19) | 0 (0) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 4 (4) | 3 (5) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 2 (5) | 8 (9) | 9 (11) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 2 (4) | 16 (22) | 7 (18) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 2 (3) | 43 (64) | 11 (14) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 9 (13) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 4 (7) | 62 (87) | 57 (86) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 23 (39) | 24 (32) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 7 (11) | 209 (398) | 195 (466) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 2 (2) | 129 (236) | 180 (353) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 148 (174) | 96 (108) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 2 (3) | 114 (233) | 93 (256) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 5 (8) | 173 (208) | 117 (153) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 21 (27) | 7 (10) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 36 (58) | 26 (37) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 56 (80) | 52 (74) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 28 (39) | 20 (28) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 71 (128) | 44 (61) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 28 (39) | 15 (20) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 34 (43) | 25 (25) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 48 (59) | 18 (18) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 36 (39) | 27 (32) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 9 (11) | 6 (6) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 27 (32) | 5 (5) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 9 (9) | 3 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 22 (22) | 26 (29) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 6 (7) | 7 (9) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 27 (29) | 41 (45) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (5) | 26 (31) | 19 (21) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 5 (6) | 73 (89) | 103 (132) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 1 (2) | 7 (12) | 17 (37) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 27 (36) | 36 (67) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 54 (61) | 81 (89) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 31 (32) | 26 (30) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 99 (188) | 6 (6) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 28 (31) | 22 (23) | 0 (0) | 0 (0)
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 24 (25) | 6 (7) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 25 (26) | 12 (12) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 23 (25) | 22 (26) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 16 (23) | 19 (25) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 12 (13) | 14 (15) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 10 (10) | 2 (2) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 (8) | 97 (114) | 60 (71) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 51 (69) | 15 (17) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 53 (67) | 17 (21) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 146 (218) | 22 (27) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 12 (12) | 12 (12) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT04662710/Prot_SAP_001.pdf